CLINICAL TRIAL: NCT00649740
Title: Single-Dose Fasting Bioequivalence Study of Topiramate Sprinkle Capsules (25 mg; Mylan) and Topamax® Sprinkle Capsules (25 mg; Ortho-McNeil Neurologics) in Healthy Volunteers
Brief Title: Fasting Study of Topiramate Sprinkle Capsules 25 mg and Topamax® Sprinkle Capsules 25 mg
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Mylan Pharmaceuticals Inc (Industry)
Responsible Party: Wayne Talton, Mylan Inc.
Organization: Viatris Inc. (Industry)
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: TOPR-0583
Record Dates: First submitted 2008-03-30; First posted 2008-04-01 (Estimated); Last update posted 2024-04-23 (Actual); Status verified 2024-04

CONDITIONS: Healthy

ARMS (2):
- 1 (Experimental): Topiramate Sprinkle Capsules 25 mg
  Interventions: Drug: Topiramate Sprinkle Capsules 25 mg
- 2 (Active Comparator): Topamax® Sprinkle Capsule 25 mg
  Interventions: Drug: Topamax® Sprinkle Capsule 25 mg

INTERVENTIONS:
Drug: Topiramate Sprinkle Capsules 25 mg — 25mg, single dose fasting
  Arms: 1
Drug: Topamax® Sprinkle Capsule 25 mg — 25mg, single dose fasting
  Arms: 2

SUMMARY:
The objective of this study was to investigate the bioequivalence of Mylan's topiramate sprinkle 25 mg capsule to Ortho-McNeil's Topamax® Sprinkle 25 mg capsule following a single, oral 25 mg (1 x 25 mg) dose administered under fasting conditions.

ELIGIBILITY:
Inclusion Criteria:

* healthy, adult subjects, 18 years and older
* able to swallow medication

Exclusion Criteria:

* institutionalized subjects
* history of any significant disease
* use of any prescription or OTC medications within 14 days of start of study
* received any investigational products within 30 days prior to start of study

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2005-11; Primary Completion 2005-12 (Actual); Study Completion 2005-12 (Actual)

PRIMARY OUTCOMES:
The 90% confidence interval for the LSMeans ratio of CPEAK, AUCL, and AUCI for the test and reference product should be between 80.00% and 125.00% for the natural log-transformed data. | blood collections through 144 hours

CONTACTS AND LOCATIONS:
Overall Officials: Dorian Williams, M.D., Principal Investigator — Kendle International Inc.
Locations (1):
- Kendle International Inc., Morgantown, West Virginia, United States

REFERENCES:
- See also: Mylan Pharmaceuticals Inc. - Clinical Trial Results — http://www.mpibiostudies.com
- See also: Daily Med - posting of most recent submitted labelling to the Food and Drug Administration (FDA) and currently in use — http://dailymed.nlm.nih.gov/dailymed/about.cfm
- See also: Recalls, Market Withdrawals and Safety Alerts — http://www.fda.gov/opacom/7alerts.html